CLINICAL TRIAL: NCT05838573
Title: The Effect of Metformin Treatment on Cognitive Impairment in Individuals With Schizophrenia: A 24-week Multicentre Randomised Controlled Trial
Brief Title: Metformin Treatment on Cognitive Impairment of Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Shandong Mental Health Center (Other); The Second People's Hospital of Dali Bai Autonomous Prefecture (Unknown); The Third people's Hospital of Jiangyin (Unknown)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WU202211MET
Record Dates: First submitted 2023-03-22; First posted 2023-05-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive impairment; Metformin; Clinical trial
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two groups were observed longitudinally for 24 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Metformin group (Active Comparator): The goal is to investigate whether adding metformin will benefit the cognitive impairment in individuals with schizophrenia.
  Interventions: Drug: Metformin treatment
- Placebo group (Placebo Comparator): The purpose of using placebo is to judge if the outcome is related to the study medication rather than other reasons.
  Interventions: Drug: Placebo treatment
- Cross-sectional participants (Experimental): Participants do not meet any of the diagnostic criteria for metabolic syndrome: 1)abdominal obesity (i.e. central obesity): waist circumference for male≥90 cm, for female ≥85 cm; 2)fasting blood glucose ≥110 mg/dl (6.1 mmol/l) and/or plasma glucose ≥140 mg/dl (7.8 mmol/l) after glucose load; 3)at fasting state, triglyceride ≥1.7 mmol/l; 4)at fasting state, HDL-C <1.04 mmol/L.
  the other inclusion criteria and exclusion criteria are same as the intervention group.
  Interventions: Other: Baseline assessments
- Healthy volunteer (Experimental)
  Interventions: Other: Volunteer assessments

INTERVENTIONS:
Drug: Metformin treatment — Participants assigned to the metformin group will receive 500mg metformin three times daily (tid) for 24 weeks. The initial dose will be 500 mg orally in the evening for the first two days, followed by an increase to 500mg twice a day for the subsequent two days. By day 5, the dosage will be further increased to 500mg tid. The highest tolerated dosage will be maintained for participants who could not tolerate the maximum dosage.
  Arms: Metformin group
Drug: Placebo treatment — Parallel-dose adjustments will be made for the placebo group to maintain consistency in dosing between the two groups.
  Arms: Placebo group
Other: Baseline assessments — Schizophrenic participants who don't meet any of the diagnostic criteria for metabolic syndrome will only accept baseline evaluations.
  Arms: Cross-sectional participants
Other: Volunteer assessments — Apart from psychiatry scales(Hamilton Depression Scale, Young Mania Rating Scale and Self-reporting Inventory-90), other assessments for the healthy subjects are the same as the baseline for sczhiophrenic participants.
  Arms: Healthy volunteer

SUMMARY:
In this study, the investigators will investigate the effect and the underlying mechanism of metformin treatment on cognitive impairment in individuals with schizophrenia. The study will recruit 120 individuals with schizophrenia at 4 sites, who will be randomized to metformin or placebo group for 24-week treatment. Clinical assessments will be done at screen/baseline, 12th week and 24th week. Participants who don't meet any of the diagnostic criteria for metabolic syndrome will only accept baseline evaluations. The specific aims are to compare healthy volunteers versus schizophrenic participants on:1) cognition; 2) MRI features, and to compare metformin group versus placebo group of 24-week treatment cohort on: 1) cognition; 2) clinical core symptoms; 3) MRI features. Biological samples also will be collected and stored to explore related mechanisms.

DETAILED DESCRIPTION:
Participants screened through inclusion and exclusion criteria will be randomized to metformin or placebo group (2:1). The information of demographic data, medical history, previous and current medication regimen, and family history regarding psychotic and metabolic diseases will be collected at baseline. The assessments will be carried out at baseline, 12th week and 24th week, including physical examination, anthropometry, blood test(blood routine, liver function, renal function, blood lipids, fasting blood glucose, serum insulin and thyroid function), electrocardiogram, MRI scan( High-resolution T1-weighted Anatomical Images, Diffusion Tensor Imaging, Resting-state functional MRI and Arterial Spin Labeling) and psychiatry scales(Positive And Negative Syndrome Scale, Scale for Assessment of Negative Symptoms, Calgary Depressing Scale for Schizophrenia, Personal and Social Performance Scale, The Systematic Assessment for Treatment Emergent Events, the Simpson-Angus Extrapyramidal Side Effects Scale and the Barnes Akathisia Rating Scale); cognitive function will be assessed by the Measurement and Treatment Research to Improve Cognition in Schizophrenia(MATRICS) Consensus Cognitive Battery; biological samples also will be collected and stored to explore related mechanisms. Participants who don't meet any of the diagnostic criteria for metabolic syndrome will only accept baseline evaluations. In addition, we will recruit healthy volunteers, and collect their demographic data, and family history regarding psychotic and metabolic diseases. Apart from psychiatry scales(Hamilton Depression Scale, Young Mania Rating Scale and Self-reporting Inventory-90), other assessments for the healthy subjects are the same as the baseline for sczhiophrenic participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 to 50 years, who meet the Diagnostic and Statistical Manual (DSM-5) diagnostic criteria for schizophrenia.
2. Duration of illness less than 15 years with current symptoms in a stable condition.
3. Participants must be receiving stable treatment with standard-of-care medications, with a maximum allowance of two antipsychotic medications. If additional anticholinergic agents are required for the management of extrapyramidal symptoms, they should be prescribed at low dosages.
4. Have great compliance with medication and follow-up.
5. Meet one of the diagnostic criteria for metabolic syndrome: 1)abdominal obesity (i.e. central obesity): waist circumference for male≥90 cm, for female ≥85 cm; 2)fasting blood glucose ≥110 mg/dl (6.1 mmol/l) and/or plasma glucose ≥140 mg/dl (7.8 mmol/l) after glucose load; 3)at fasting state, triglyceride ≥1.7 mmol/l; 4)at fasting state, HDL-C <1.04 mmol/L.
6. Signed the study consent for participation.

Exclusion Criteria:

1. Having a history of substance dependence or abuse or whose symptoms are caused by other diagnosable mental disorders.
2. Having a history of traumatic brain injury, seizures or other known neurological or organic diseases of the central nervous system.
3. Taking antidepressants, stimulants, mood stabilizers or accepts electricity shock treatment.
4. Having current suicidal or homicidal thoughts or any safety concern by research staff that cannot be managed in an inpatient setting.
5. Taking dementia related drugs, minocycline, and other drugs that could affect cognitive function.
6. The routine blood tests showing significant abnormal renal, liver function or other somatic disease.
7. Pregnant or lactating women.

For schizophrenic participants who don't meet any of the diagnostic criteria for metabolic syndrome will only accept baseline evaluations.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of the score of the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery of interventional participants | From baseline to 12th week；From baseline to 24th week；
  At baseline and 12th week, the cognitive function of interventional participants will be assessed using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery. Evaluator convert raw scores to scale scores, then to normalized T scores. T scores of seven domains and composite score are further calculated. The changes of scores after 12-week metformin treatment will be used for assessing the improvement of cognitive function (higher score means better function).
Changes of brain cerebral blood flow by arterial spin labeling of interventional participants | From baseline to 12th week；From baseline to 24th week
  At baseline and 12th week, whole brain cerebral blood flow (CBF) will be recorded by arterial spin labeling (ASL). For interventional participants, the changes in CBF (c-CBF) before and after the application of 160 units nasal insulin spray of interventional participants will be calculated. The changes of c-CBF after 12-week metformin treatment will be reported.

SECONDARY OUTCOMES:
Changes of resting-state functional MRI of interventional participants | From baseline to 12th week; From baseline to 24th week
  At each visit, the resting-state functional MRI(fMRI) will be conducted at fasting state. For interventional participants, the changes in fMRI (c-fMRI) before and after the application of 160 units nasal insulin spray will be analysed. The changes of c-fMRI after 24-week metformin treatment will be used for exploring underlying mechanism.
Changes of social function by Personal and Social Performance Scale | From baseline to 24th week
  The changes of Personal and Social Performance Scale of interventional participants at different follow up timepoint will be used for evaluating the improvement of personal life and social function.(higher score means better function)
Changes of clinical symptoms by Scale for Assessment of Negative Symptoms | From baseline to 24th week
  The changes of Scale for Assessment of Negative Symptoms of interventional participants at different follow up timepoint will be used for recording the improvement of negative symptoms.(lower score means alleviation of symptoms)
Changes of clinical symptoms by Positive And Negative Syndrome Scale | From baseline to 24th week
  The changes of Positive And Negative Syndrome Scale of interventional participants at different follow up timepoint will be used for recording the improvement of psychiatric symptoms.(lower score means alleviation of symptoms)
Changes of homoeostasis model assessment-estimated insulin resistance | From baseline to 24th week
  Homoeostasis model assessment-estimated insulin resistance (HOMA-IR) represents systemic insulin resistance(higher value means worse outcome). For interventional participants, the changes of HOMA-IR will partly reflect the changes of peripheral insulin resistance after metfromin treament.
The difference of cerebral blood flow between schizophrenic participants and healthy volunteers | Baseline
  At baseline, whole brain cerebral blood flow (CBF) will be recorded by arterial spin labeling (ASL) for every participants, the changes in CBF (c-CBF) before and after the application of 160 units nasal insulin spray will be calculated. The difference of c-CBF of the brain between schizophrenic participants and healthy volunteers will be reported.
The difference of resting-state functional MRI between schizophrenic participants and healthy volunteers | Baseline
  At baseline, the resting-state functional MRI(fMRI) will be conducted at fasting state. For every participants, the changes in fMRI (c-fMRI) before and after the application of 160 units nasal insulin spray will be analysed. The c-fMRI between schizophrenic participants and healthy volunteers may reflect the underlying mechanism of disease.
The difference of the score of the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery between schizophrenic participants and healthy volunteers | Baseline
  At baseline, the cognitive function will be assessed using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery, including schizophrenic participants and healthy volunteers. Evaluator convert raw scores to scale scores, then to normalized T scores. T scores of seven domains and composite score are further calculated(higher score means better function). The difference of scores and their relationships with cerebral blood flow (CBF) and resting-state functional MRI(fMRI) will be used for exploring underlying mechanism.

OTHER OUTCOMES:
High-resolution T1-weighted anatomical images and Diffusion Tensor Imaging by MRI at baseline for predicting efficacy | From baseline to 24th week
  T1-weighted images will be acquired using 3D inversion recovery-prepared fast spoiled gradient-echo sequences, while Diffusion Tensor Imaging (DTI) will be performed using diffusion-weighted echo planar imaging sequences. The T1-weighted mages and DTI acquired at baseline will be analysed for predicting efficacy of metformin on cognitive function for interventional participants.
The difference of Diffusion Tensor Imaging scanned by MRI between schizophrenic participants and healthy volunteers | Baseline
  Diffusion Tensor Imaging (DTI) will be performed using diffusion-weighted echo planar imaging sequences. The analysis of DTI will be conducted to investigate the difference of brain structure and morphology between schizophrenic participants and healthy volunteers.
Safety evaluation through the Systematic Assessment for Treatment Emergent Events | From baseline to 24th week
  The participants will be asked to score the occurred side effects using the Systematic Assessment for Treatment Emergent Events at every visit. (higher score means worse side effect)

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, M.D., Ph.D., Study Chair — Mental Health Institute of Second Xiangya Hospital,CSU
Locations (4):
- China (4):
  - Mental Health Institute of Second Xiangya Hospital,CSU, Changsha, Hunan
  - The Third Peoples's Hospital of Jiangyin, Jiangyin, Jiangsu
  - Shandong Mental Health Center, Jinan, Shandong
  - The Second People's Hospital of Dali Bai Autonomous Prefecture, Dali, Yunnan

IPD SHARING:
Plan to Share IPD: No